CLINICAL TRIAL: NCT01624259
Title: A Randomized, Open-Label, Parallel-Arm Study Comparing the Effect of Once-Weekly Dulaglutide With Once-Daily Liraglutide in Patients With Type 2 Diabetes (AWARD-6: Assessment of Weekly AdministRation of LY2189265 in Diabetes-6)
Brief Title: A Study Comparing the Effect of Dulaglutide With Liraglutide in Type 2 Diabetes
Acronym: AWARD-6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11377; H9X-MC-GBDE (Other: Eli Lilly and Company); 2011-003810-18 (EudraCT Number)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 26 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
  Interventions: Drug: LY2189265; Drug: Metformin
- Liraglutide (Active Comparator): Liraglutide 0.6 mg, SC, once daily for 7 days, then titrated up to Liraglutide 1.2 mg, SC, once daily for 7 days, then titrated up to Liraglutide 1.8 mg, SC, once daily for 24 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: LY2189265 — Administered SC
  Other Names: Dulaglutide
  Arms: 1.5 mg LY2189265
Drug: Liraglutide — Administered SC
  Arms: Liraglutide
Drug: Metformin

SUMMARY:
The purpose of the study is to assess the benefits and risks of once-weekly dulaglutide compared to once-daily liraglutide in participants with type 2 diabetes who have inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Not optimally controlled on diet and exercise and a dose of metformin that is at least 1500 milligrams/day (mg/day) and has been at a stable dose for at least 3 months prior to the first study visit
* Glycosylated hemoglobin (HbA1c) greater than or equal to 7.0% and less than or equal to 10.0%
* Accept continued treatment with metformin throughout the trial, as required per protocol
* Men and nonpregnant women aged greater than or equal to 18 years
* Stable weight (plus or minus 5%) greater than or equal to 3 months prior to screening
* Body Mass Index (BMI) less than or equal to 45 kilograms/square meter (kg/m^2)

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have been treated with ANY other antihyperglycemic medications (other than metformin) at the time of the first study visit or within the 3 months prior to the first study visit
* Have used insulin therapy (outside of pregnancy) any time in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 weeks; any insulin use within 3 months prior to the first study visit
* Have been treated with drugs that promote weight loss within 3 months of the first study visit
* Are receiving chronic (greater than 14 days) systemic glucocorticoid therapy or have received such therapy within the 4 weeks immediately prior to the first study visit
* Have had any of the following cardiovascular conditions within 2 months prior to the first study visit: acute myocardial infarction, New York Heart Association Class III or Class IV heart failure, or cerebrovascular accident
* Have a known clinically significant gastric emptying abnormality (such as, severe diabetic gastroparesis or gastric outlet obstruction) or have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or alanine transaminase level greater than or equal to 3 times the upper limit of normal
* Have a history of chronic pancreatitis or acute idiopathic pancreatitis or were diagnosed with any type of acute pancreatitis within the 3 month period prior to the first study visit
* Have a serum creatinine greater than or equal to 1.5 milligrams/deciliter (mg/dL) (male) or greater than or equal to 1.4 mg/dL (female), or a creatinine clearance less than 60 milliliters/minute (mL/minute)
* Have any self or family history of type 2A or type 2B multiple endocrine neoplasia (MEN 2A or 2B, respectively) in the absence of known C-cell hyperplasia (this exclusion includes those participants with a family history of MEN 2A or 2B whose family history for the syndrome is Rearranged during Transfection (RET) negative; the only exception for this exclusion will be for participants whose family members with MEN 2A or 2B have a known RET mutation and the potential participant for the study is negative for that RET mutation)
* Have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, or carcinoma (including sporadic, familial, or part of MEN 2A or 2B syndrome)
* Have a serum calcitonin greater than or equal to 20 picograms/milliliter (pg/mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (57):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perrysburg, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingsport, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hurst, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hohenmölsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neunkirchen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Ingbert-Oberwürzbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sulzbach
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dombóvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey, Mexico
- Poland (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kamieniec Ząbkowicki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ruda Śląska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tychy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Río Grande
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sibiu
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malacky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nitra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nové Mesto nad Váhom
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Centelles
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrel

REFERENCES:
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396
- [Derived] Dungan KM, Povedano ST, Forst T, Gonzalez JG, Atisso C, Sealls W, Fahrbach JL. Once-weekly dulaglutide versus once-daily liraglutide in metformin-treated patients with type 2 diabetes (AWARD-6): a randomised, open-label, phase 3, non-inferiority trial. Lancet. 2014 Oct 11;384(9951):1349-57. doi: 10.1016/S0140-6736(14)60976-4. Epub 2014 Jul 10. PMID 25018121

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265: LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 26 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
- Liraglutide: Liraglutide: 0.6 mg, SC, once daily for 7 days, then titrated up to 1.2 mg, SC, once daily for 7 days, then titrated up to 1.8 mg, SC, once daily for 24 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
Period: Overall Study
Arm/Group | LY2189265 | Liraglutide
Started | 299 | 300
Received at Least One Dose of Study Drug | 299 | 300
Completed | 269 (Completed the study on study treatment) | 269 (Completed the study on study treatment)
Not Completed | 30 | 31
Not completed — Adverse Event | 18 | 18
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Abnormal laboratory measure | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide
Groups:
- LY2189265: LY2189265 (Dulaglutide): 1.5 mg, SC, once weekly for 26 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
- Liraglutide: Liraglutide 0.6 mg, SC, once daily for 7 days, then titrated up to 1.2 mg, SC, once daily for 7 days, then titrated up to 1.8 mg, SC, once daily for 24 weeks
  Metformin: at least 1500 mg/day, oral, for 26 weeks
- Total: Total of all reporting groups
Arm/Group | LY2189265 | Liraglutide | Total
Number analyzed (Participants) | 299 | 300 | 599
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.49 (9.34) | 56.81 (9.91) | 56.65 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 151 | 312
  Male | 138 | 149 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 72 | 147
  Not Hispanic or Latino | 221 | 223 | 444
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 23 | 43
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 16 | 37
  White | 256 | 259 | 515
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 97 | 97 | 194
  Czech Republic | 27 | 28 | 55
  Hungary | 21 | 19 | 40
  Mexico | 20 | 21 | 41
  Slovakia | 20 | 22 | 42
  Puerto Rico | 3 | 4 | 7
  Poland | 39 | 42 | 81
  Spain | 24 | 24 | 48
  Romania | 20 | 17 | 37
  Germany | 28 | 26 | 54
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 93.82 (18.23) | 94.35 (18.96) | 94.09 (18.58)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared
  kilograms per meter squared (kg/m^2) | 33.50 (5.07) | 33.62 (5.16) | 33.56 (5.11)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.06 (0.81) | 8.05 (0.79) | 8.05 (0.80)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 7.13 (5.41) | 7.28 (5.41) | 7.21 (5.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26 Weeks Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means of the glycosylated hemoglobin A1c (HbA1c) change from baseline to the primary endpoint at Week 26 was adjusted by fixed effects of treatment, country, visit, treatment-by-visit interaction, participant as random effect, and baseline HbA1c as covariates, via a mixed-effects model for repeated measures (MMRM) analysis using restricted maximum likelihood (REML).
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide with evaluable HbA1c data
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- 1.5 mg LY2189265: LY2189265 (Dulaglutide): 1.5 mg, SC, once weekly for 26 weeks
  Metformin: at least 1500 mg/day, administered orally, for 26 weeks
- 1.8 mg Liraglutide: Liraglutide: 0.6 mg, SC, once daily for 7 days, then titrated up to 1.2 mg, SC, once daily for 7 days, then titrated up to 1.8 mg, SC, once daily for 24 weeks
  Metformin: at least 1500 mg/day, administered orally, for 26 weeks
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 279 | 272
percentage of glycosylated hemoglobin | -1.42 (0.05) | -1.36 (0.05)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; To show noninferiority of 1.5 mg LY2189265 relative to 1.8 mg liraglutide with 90% power, 222 completers (444 total) at 26 weeks were required. Noninferiority of 1.5 mg LY2189265 relative to 1.8 mg liraglutide was demonstrated if the upper bound of the two-sided 95% Confidence Interval (CI) for the difference in mean change in HbA1c between the 1.5 mg LY2189265 arm and 1.8 mg liraglutide arm was below 0.4%; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying a serial gatekeeping strategy. This calculation assumed a 0 difference in HbA1c between the 1.5 mg LY2189265 1.5-mg arm and 1.8 mg liraglutide, 0.4% margin of noninferiority, common Standard Deviation (SD) of 1.3% for change from baseline in HbA1c, 0.05 two-sided significance level, and 25% dropout rate at 26 weeks; p < 0.001, Mixed Models Analysis — 1-sided raw p-value (no multiplicity adjustment); LS Mean Difference = -0.06, 95% CI 2-sided [-0.19 to 0.07]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Superiority analysis; Test type: Superiority or Other; p = 0.186, Mixed Models Analysis — 1-sided raw p-value (no multiplicity adjustment); LS Mean Difference = -0.06, 95% CI 2-sided [-0.19 to 0.07]

2. Secondary Outcome: Change From Baseline in Body Weight at 26 Weeks
Description: LS means of the weight change from baseline to primary endpoint at Week 26 were calculated using analysis of covariance (ANCOVA) with HbA1c Strata, country, and treatment as fixed effects and baseline body weight as a covariate.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide with evaluable body weight data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 299
kilograms (kg) | -2.90 (0.22) | -3.61 (0.22)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Treatment comparison from ANCOVA model at 26 weeks; Test type: Superiority or Other; p = 0.010, ANCOVA — No adjustment for multiplicity; LS Mean Difference = 0.71, 95% CI 2-sided [0.17 to 1.26], Standard Error of Mean 0.28

3. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at 26 Weeks
Description: BMI is an estimate of body fat based on body weight divided by height squared. LS means of the BMI change from baseline to primary endpoint at Week 26 were calculated using ANCOVA with HbA1c Strata, country, and treatment as fixed effects and baseline BMI as a covariate.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable BMI data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms/square meter (kg/m^2)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 299
kilograms/square meter (kg/m^2) | -1.05 (0.08) | -1.30 (0.08)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Treatment comparison from ANCOVA model; Test type: Superiority or Other; p = 0.013, ANCOVA — No adjustment for multiplicity; LS Mean Difference = 0.25, 95% CI 2-sided [0.05 to 0.45], Standard Error of Mean 0.10

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 26 Weeks
Description: LS means of the FPG from baseline to primary endpoint at Week 26 were adjusted by fixed effects of treatment, country, baseline HbA1c strata, and baseline FPG as covariates, via ANCOVA with LOCF.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable FPG data. Only pre-rescue measurements were used.
  LOCF was used to impute missing postbaseline values. If no data after date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 281 | 277
milligrams/deciliter (mg/dL) | -34.81 (2.13) | -34.25 (2.11)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Treatment comparison from ANCOVA model; Test type: Superiority or Other; p = 0.828, ANCOVA — No adjustment for multiplicity; LS Mean Difference = -0.57, 95% CI 2-sided [-5.69 to 4.56], Standard Error of Mean 2.61

5. Secondary Outcome: Change From Baseline in 7-Point Self Monitored Plasma Glucose (SMPG) at 26 Weeks
Description: The SMPG data were collected at the following 7 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening meal; 2 hours post-evening meal; and bedtime. The mean of the 7 time points (Daily Mean) was also calculated.
  LS means of the SMPG change from baseline to primary endpoint at Week 26 were adjusted by fixed effects of treatment, HbA1c strata, country, visit, treatment-by-visit interaction, participant as random effect and baseline SMPG as a covariate, via a MMRM analysis using REML.
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable 7-Point SMPG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 248 | 256
mg/dL | -40.76 (1.50) | -38.51 (1.45)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Test type: Superiority or Other; p = 0.228, Mixed Models Analysis — No adjustment for multiplicity; P-value from pairwise comparison of LS means at 26 weeks from REML-based MMRM; LS Mean Difference = -2.25, 95% CI 2-sided [-5.91 to 1.41], Standard Error of Mean 1.86

6. Secondary Outcome: Percentage of Participants Achieving a Glycosylated Hemoglobin (HbA1c) ≤6.5% or <7% at 26 Weeks
Description: The percentage of participants who achieved the target HbA1c values at the primary endpoint were analyzed with a repeated logistic regression model (the generalized estimation equation [GEE] model). The model includes pooled country, treatment, visit, treatment-by-visit interaction, and baseline HbA1c as continuous covariates.
Time Frame: Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide with evaluable HbA1c data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 293 | 293
percentage of participants
  HbA1c levels ≤6.5% | 54.6 | 50.9
  HbA1c levels <7.0% | 68.3 | 67.9
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Treatment comparison for HbA1c levels ≤6.5%; Test type: Superiority or Other; p = 0.322, Regression, Logistic — P-value of treatment comparison at Week 26 is from repeated generalized linear mixed model (GLM model); No adjustment for multiplicity; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.81 to 1.86]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Treatment comparison for HbA1c levels <7.0%; Test type: Superiority or Other; p = 0.925, Regression, Logistic — No adjustment for multiplicity; P-value of treatment comparison at Week 26 is from repeated generalized linear mixed model (GLM model); Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.64 to 1.63]

7. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Steady-state Beta (β)- Cell Function (HOMA2-%B) at 26 Weeks
Description: The homeostatic model assessment (HOMA) quantifies insulin resistance and beta-cell function. HOMA2-%B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady-state beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%.
  LS means of the HOMA2-%B change from baseline to primary endpoint at Week 26 was adjusted by fixed effects of treatment, country, baseline HbA1c strata, and baseline HOMA2-%B value as covariate, via an ANCOVA analysis using LOCF.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable HOMA2-%B data. LOCF was used to impute missing postbaseline values. If there was no data after date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%B
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 275 | 265
percentage of HOMA2-%B | 37.03 (2.26) | 35.59 (2.27)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs 1.8 mg Liraglutide; Test type: Superiority or Other; p = 0.608, ANCOVA; No adjustment for multiplicity; LS Mean Difference = 1.43, 95% CI 2-sided [-4.06 to 6.92], Standard Error of Mean 2.79

8. Secondary Outcome: Number of Participants With Reported and Adjudicated Cardiovascular Events
Description: Deaths and nonfatal cardiovascular (CV) adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal CV AEs to be adjudicated include myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with reported CV events, number of participants with nonfatal CV events confirmed by adjudication, and number of deaths confirmed by adjudication are summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable adjudicated CV event data.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
participants
  Any reported CV events | 0 | 3
  Any adjudicated nonfatal CV events | 0 | 1
  Any confirmed adjudicated deaths | 0 | 0

9. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters, Heart Rate (HR) at 26 Weeks
Description: ECG HR was measured. LS means of change from baseline were analyzed using ANCOVA with HbA1c strata, country, and treatment as fixed effects and baseline HR as a covariate.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable ECG heart rate data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 273 | 284
beats per minute (bpm) | 1.9 (0.55) | 4.1 (0.54)

10. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters PR and QTcF (Fridericia's) Intervals at 26 Weeks
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave. QTcF is the measure of the time between the start of the Q wave and the end of the T wave adjusted using Fridericia's formula. PR is the interval between the P wave and the QRS complex. These parameters were calculated from electrocardiogram (ECG) data. LS means of change from baseline for the PR and QTcF intervals will be analyzed using the MMRM similar to MMRM model for primary outcome, using corresponding baseline and HbA1c strata. Only ECGs obtained at scheduled visits will be used in these summaries and analyses.
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide with evaluable ECG PR or QTcF interval data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 273 | 284
milliseconds (msec)
  PR interval (n=270, 278) | 3.8 (0.81) | 3.3 (0.80)
  QTcF interval (n=273, 284) | 0.39 (0.90) | -0.72 (0.89)

11. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 26 Weeks
Description: Descriptive statistics for the actual measurements and LS means of change from baseline for HR (sitting) by treatment arm were analyzed using the MMRM model with treatment, country, visit, and treatment-by-visit interaction as fixed effects, baseline rate as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable heart rate data.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 288 | 288
bpm | 2.37 (0.4) | 3.12 (0.4)

12. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at 26 Weeks
Description: Descriptive statistics for the actual measurements and change from baseline for sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured. LS means of change from baseline were calculated using MMRM with treatment, country, visit, and treatment-by-visit interaction as fixed effects, baseline BP as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable BP data.
Measure: Least Squares Mean (Standard Error); unit: milliliters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 278 | 281
milliliters of mercury (mmHg)
  Sitting DBP | -0.22 (0.4) | -0.31 (0.4)
  Sitting SBP | -3.36 (0.7) | -2.82 (0.7)

13. Secondary Outcome: Number of Participants With Adjudicated Acute Pancreatitis Events
Description: The number of participants with events of pancreatitis confirmed by adjudication were summarized cumulatively at 26 weeks (including a 30-day follow up). Pancreatitis events were adjudicated by a committee of physicians external to the Sponsor.
  A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to 30 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Liraglutide with evaluable adverse event data.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
participants | 0 | 0

14. Secondary Outcome: Change From Baseline in Calcitonin at 26 Weeks
Description: A summary of participants having changes in calcitonin values from baseline to primary endpoint of 26 weeks is presented.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable calcitonin laboratory data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: picograms/milliliter (pcg/mL)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 292 | 294
picograms/milliliter (pcg/mL) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

15. Secondary Outcome: Change From Baseline in Lipase at 26 Weeks
Description: A summary of participants having changes in lipase evaluation from baseline to primary endpoint of 26 weeks is presented.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable lipase laboratory data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units/liter (U/L)
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 288 | 289
units/liter (U/L) | 7.0 [0.5 to 17.5] | 11.0 [2.0 to 23.0]

16. Secondary Outcome: Change From Baseline in Amylase at 26 Weeks
Description: A summary of participants having changes in amylase evaluation from baseline to primary endpoint of 26 weeks is presented.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable amylase laboratory data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 287 | 289
U/L | 7.0 [0.0 to 14.0] | 6.0 [0.0 to 13.0]

17. Secondary Outcome: Percentage of Participants With Self-Reported Hypoglycemia Events
Description: Hypoglycemic events (HE) were classified as severe (episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (any time a participant felt that he/she was experiencing symptoms and/or signs associated with hypoglycemia and had a plasma glucose [PG] concentration of ≤70 mg/dL), asymptomatic (events not accompanied by typical symptoms of hypoglycemia but with a measured PG of ≤ 70 mg/dL), nocturnal (events that occurred between bedtime and waking), or probable symptomatic (events during which symptoms of hypoglycemia were not accompanied by a PG determination but that was presumably caused by a PG of ≤70 mg/dL).
  A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable hypoglycemia event data. Only pre-rescue measurements were used.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
percentage of participants
  Documented symptomatic HE | 2.7 | 2.7
  Asymptomatic HE | 6.7 | 3.3
  Severe HE | 0.0 | 0.0
  Nocturnal HE | 1.3 | 2.0
  Probable symptomatic HE | 1.0 | 1.0

18. Secondary Outcome: Percentage of Participants Requiring Additional Intervention for Severe, Persistent Hyperglycemia
Description: An additional intervention (rescue therapy) was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation.
Time Frame: Baseline through 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable concomitant medication data.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
percentage of participants | 0.3 | 1.0

19. Secondary Outcome: Rate of Hypoglycemic Events Adjusted Per 30 Days
Description: HE were classified as severe (episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (any time a participant felt that he/she was experiencing symptoms and/or signs associated with hypoglycemia and had a PG concentration of ≤70 mg/dL), asymptomatic (events not accompanied by typical symptoms of hypoglycemia but with a measured PG of ≤ 70 mg/dL), nocturnal (events that occurred between bedtime and waking), or probable symptomatic (events during which symptoms of hypoglycemia were not accompanied by a PG determination but that was presumably caused by a PG of ≤70 mg/dL). The hypoglycemia rate per 30 days was calculated by the number of hypoglycemia events within the period/number of days participant at risk within the period*30 days. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable hypoglycemic episode data. Only pre-rescue measurements were used.
Measure: Mean (Standard Deviation); unit: number of events/participant/30 days
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
number of events/participant/30 days
  Total HE | 0.03 (0.12) | 0.04 (0.25)
  Documented symptomatic HE | 0.01 (0.08) | 0.02 (0.17)
  Asymptomatic HE | 0.02 (0.07) | 0.01 (0.08)
  Severe HE | 0.00 (0.00) | 0.00 (0.00)
  Nocturnal HE | 0.01 (0.05) | 0.01 (0.10)
  Probable symptomatic HE | 0.00 (0.02) | 0.01 (1.12)

20. Secondary Outcome: Time to Initiation of Additional Intervention for Severe, Persistent Hyperglycemia
Description: An additional intervention (rescue therapy) was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. Participants who had no rescue therapy within specified study period were considered as censored observations at the last available contact date up to specified study period.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
weeks | NA [0.975 to 1.000] — A median time to initiation of additional intervention could not be calculated due to the small number of events requiring rescue therapy. | NA [0.966 to 0.996] — A median time to initiation of additional intervention could not be calculated due to the small number of events requiring rescue therapy.

21. Secondary Outcome: Number of Participants With Allergic or Hypersensitivity Reactions
Description: Allergic and hypersensitivity reactions that were considered possibly related to study drug by the investigator are presented. Serious and all other non-serious adverse events regardless of causality are summarized in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Number analyzed (Participants) | 299 | 300
participants | 1 | 5

22. Secondary Outcome: Number of Participants With Treatment Emergent LY2189265 Antibodies up to 26 Weeks and 4 Weeks After Last Dose
Description: LY2189265 (dulaglutide) anti-drug antibodies (ADA) were assessed at baseline, 26 weeks, and at the safety follow-up visit 4 weeks after study drug discontinuation in dulaglutide-treated participants. A participant was considered to have treatment emergent LY2189265 ADA if the participant had at least 1 titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement. The number of participants with treatment-emergent LY2189265 ADA from postbaseline to follow up were summarized.
Time Frame: Baseline up to 4 Weeks Post Last Dose of Study Drug
Population: Participants who were randomized and received at least 1 dose of LY2189265 with evaluable LY2189265 ADA data.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265
Number analyzed (Participants) | 290
participants | 3

23. Secondary Outcome: Percent Change From Baseline in Lipid Parameters at 26 Weeks
Description: A summary of percent change in lipid parameters (total cholesterol, high-density lipoprotein cholesterol [HDL-C], low density lipoprotein cholesterol [LDL-C], very low-density lipoprotein cholesterol [VLDL], and triglycerides) from baseline to primary endpoint of 26 weeks is presented. LS means of the lipid parameter from baseline to primary endpoint at Week 26 were adjusted by fixed effects of treatment, country, baseline HbA1c strata, and lipid parameter baseline as covariates, via ANCOVA with LOCF.
Time Frame: Baseline, Up to 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or liraglutide with evaluable lipid laboratory data. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | LY2189265 | Liraglutide
Number analyzed (Participants) | 286 | 284
percent
  Total cholesterol (n=286, 284) | -1.64 (1.18) | 0.67 (1.18)
  HDL-C (n=286, 284) | 6.21 (1.02) | 6.46 (1.02)
  LDL-C (n=276, 276) | -1.09 (2.17) | 3.20 (2.15)
  VLDL (n=276, 276) | 1.56 (2.63) | 2.92 (2.60)
  Triglycerides (n=286, 284) | 0.59 (2.76) | 1.35 (2.76)

ADVERSE EVENTS:
Arm/Group | 1.5 mg LY2189265 | 1.8 mg Liraglutide
Serious Adverse Events (participants affected / at risk) | 5/299 | 11/300
Other Adverse Events (participants affected / at risk) | 185/299 | 186/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=299) | 1.8 mg Liraglutide (N=300)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (2)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=299) | 1.8 mg Liraglutide (N=300)
Constipation (Gastrointestinal disorders) | 11 (16) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 36 (56) | 36 (51)
Dyspepsia (Gastrointestinal disorders) | 24 (36) | 18 (22)
Nausea (Gastrointestinal disorders) | 61 (108) | 54 (77)
Vomiting (Gastrointestinal disorders) | 21 (24) | 25 (36)
Nasopharyngitis (Infections and infestations) | 23 (30) | 21 (24)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 20 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 15 (27)
Headache (Nervous system disorders) | 22 (36) | 25 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days